CLINICAL TRIAL: NCT00064389
Title: Long Term Safety Study of Levalbuterol and Racemic Albuterol in Subjects Twelve Years of Age and Older With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 051-356
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): levalbuterol 90 mcg MDI QID
  Interventions: Drug: levalbuterol tartrate HFA MDI
- 2 (Active Comparator): racemic albuterol HFA MDI 180 mcg QID
  Interventions: Drug: racemic albuterol

INTERVENTIONS:
Drug: levalbuterol tartrate HFA MDI — levalbuterol MDI 90 mcg QID
  Other Names: Xopenex HFA MDI
  Arms: 1
Drug: racemic albuterol — racemic albuterol HFA MDI 180 mcg QID
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety of levalbuterol as compared to racemic albuterol based on the frequencies of adverse events reporting during a 12-month period of chronic dosing of adolescent and adult subjects with asthma.

DETAILED DESCRIPTION:
This was a randomized, open-label, active controlled, multicenter, parallel-group safety study in subjects 12 years of age and older with asthma. Subjects of appropriate age who completed the Phase III levalbuterol HFA MDI trials (Studies 051-353 or 051-355) were eligible to participate. Studies 051-353 and 051-355, both entitled "An Efficacy and Safety Study of Levalbuterol, Racemic Albuterol and Placebo in Subjects Twelve Years of Age and Older with Asthma" were multicenter, randomized, double-blind, placebo- and active-controlled, parallel-group studies of up to nine weeks in duration (a one-week single-blind placebo run in period followed by an eight-week double-blind treatment period). Subjects who completed Studies 051 353 and 051 355 but who were not immediately eligible to rollover into the current study could also participate but only after a 30-day washout. New subjects and subjects who participated in the Phase III trials who were not immediately eligible (ie, had a >30-day washout) were considered to be de novo subjects.Study participation included 10 study visits over a 12 month period.

This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria

* Willing and able to comply with study procedures and visit schedules
* Females 12-60 yrs must have a negative serum pregnancy test at study start
* Women of child bearing potential must use acceptable method of birth control throughout study
* Confirmed diagnosis of asthma minimum of 6 mos. prior to study start
* Have stable baseline asthma and have been using B-adrenergic agonist, and/or anti-asthma anti-inflammatory meds, and/or OTC asthma meds. >6 mos. prior to study start
* In good health with exception of reversible airways disease and not suffering from any chronic condition that might affect their respiratory function
* Had chest X-ray w/in 12 mos. prior to randomization that is not diagnostic of pneumonia, atelectasis, pulmonary fibrotic disease, pneumothorax, chronic obstructive pulmonary disease etc.
* Subject rolling over from either Sepracor study 051-353 or 051-355 must have successfully completed the study
* Subject who is not immediately rolled over from Sepracor study 051-353 or 051-355 must wait >30 days and will be regarded as a de novo subject
* Able to complete daily diary cards and medical event calendars reliably, understand dosing instructions, demonstrate how to use the MiniWright PEF meter. Minor subjects must have a parent/legal guardian assist them during the study with these activities

Exclusion Criteria

* Female who is pregnant or lactating
* Participated in investigational drug study w/in 30 days prior to study start, or currently participating in another clinical trial, other than Sepracor studies 051-353 or 051-355
* Subject who early terminated from Sepracor study 051-353 or 051-355
* Subject whose schedule prevents him or her from taking the first daily dose of study medication and/or starting study visits before 10 AM
* Have travel commitments during the study that would interfere with trial measurements and/or compliance
* History of hospitalization for asthma w/in 45 days prior to study start, or scheduled for in-patient hospitalization, including elective surgery during the trial
* Subject with a known sensitivity to levalbuterol or racemic albuterol, or any of the excipients contained in any of these formulations
* Subject using any prescription drug with which albuterol sulfate is contraindicated
* Subject with currently diagnosed life-threatening asthma
* History of cancer (exception: basal cell carcinoma in remission)
* Subject with hyperthyroidism, diabetes, hypertension, cardiac diseases or seizure disorders that currently are not well controlled by medication or may interfere with the successful completion of this protocol
* History of substance abuse or drug abuse within 12 months preceding V1
* Subject with >10 pack/yr history of cigarette smoking or use of any tobacco products within 6 months of study start
* Documented history of bronchopulmonary aspergillosis or any form of allergic alveolitis
* Have suffered from a clinically significant upper or lower respiratory tract infection in the 2 weeks prior to study start
* Subject who is a staff member or relative of a staff member

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2003-01; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
incidence of post-randomization adverse events | Weeks -1, 0, 1, 2, 3, 10, 11, 18, 19, 22, 23, 26, 27, 30, 31, 34, 35, 38, 39, 43, 44, 47, 48, 52, 53

SECONDARY OUTCOMES:
rate of discontinuations due to adverse events | Weeks -1, 0, 1, 2, 3, 10, 11, 18, 19, 22, 23, 26, 27, 30, 31, 34, 35, 38, 39, 43, 44, 47, 48, 52, 53
time-to-selected adverse events (AEs with an incidence ≥5%) | Weeks -1, 0, 1, 2, 3, 10, 11, 18, 19, 22, 23, 26, 27, 30, 31, 34, 35, 38, 39, 43, 44, 47, 48, 52, 53
asthma attacks, asthma adverse events, and expanded-definition asthma events | Weeks -1, 0, 1, 2, 3, 10, 11, 18, 19, 22, 23, 26, 27, 30, 31, 34, 35, 38, 39, 43, 44, 47, 48, 52, 53
clinical laboratory values | Weeks -1, 0, 10, 11, 26, 27, 43, 44, 52, 53
vital signs (blood pressure, heart rate, respiration rate, and body temperature) | Weeks -1, 0, 1, 2, 3, 10, 11, 18, 19, 26, 27, 34, 35, 43, 44, 52, 53
ECG parameters | Weeks -1, 0, 1, 10, 11, 26, 27, 43, 44, 52, 53
physical examinations | Weeks -1, 0, 26, 27, 52, 53
rescue medication, and daytime asthma control days | Weeks -1, 0, 1, 2, 3, 10, 11, 18, 19, 22, 23, 26, 27, 30, 31, 34, 35, 38, 39, 43, 44, 47, 48, 52, 53
FEV1, FVC, FEF25-75%, peak expiratory flow | Weeks -1, 0, 1, 2, 3, 10, 11, 18, 19, 26, 27, 34, 35, 43, 44, 52, 53
Asthma Quality of Life Questionnaire (AQLQ) | Weeks 0, 26, 27, 52, 53
subject and physician global evaluations | Weeks 26, 27, 52, 53
(S) and (R) albuterol plasma concentrations | Weeks -1, 0, 10, 11, 26, 27, 43, 44, 52, 53
subject assessment of study inhaler device performance | Weeks -1, 0, 1, 2, 3, 10, 11, 18, 19, 22, 23, 26, 27, 30, 31, 34, 35, 38, 39, 43, 44, 47, 48, 52, 53

CONTACTS AND LOCATIONS:
Locations (96):
- United States (91):
  - Jefferson Clinic PC, Birmington, Alabama
  - Pulmonary Associates Research Division, Mobile, Alabama
  - Montgomery Pulmonary Consultants, Montgomery, Alabama
  - Center of Research Excellence, LLC, Oxford, Alabama
  - Lovelace Scientific Resources, Phoenix, Arizona
  - Alta Clinical Research, LLC, Tucson, Arizona
  - Integrated Research Group, Corona, California
  - Northern California Research Corp, Fair Oaks, California
  - Allergy, Asthma & Respiratory Care Center, Long Beach, California
  - Madera Family Medical Group, Madera, California
  - Clinical Trials of Orange County, Inc., Orange, California
  - Institute of Healthcare Assessment, Inc., San Diego, California
  - Westlake Medical Research, Inc., Westlake Village, California
  - Office of Constantine Falliers, MD, Denver, Colorado
  - Office of Gary Richmond, MD, Fort Lauderdale, Florida
  - CNS Clinical Trials, Fort Myers, Florida
  - FPA Clinical Research, Kissimmee, Florida
  - Orlando Clinic for Asthma & Respiratory Diseases, Longwood, Florida
  - Allergy Sinus Asthma Research Institute, Miami, Florida
  - Florida Center for Alergy & Asthma Research, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Family Allergy & Asthma Center, PC, Atlanta, Georgia
  - The Allergy & Asthma Clinic Research Center, Conyers, Georgia
  - Aeroallergy Research, Savannah, Georgia
  - Sneeze, Wheeze and Itch, LLC, Bloomington, Illinois
  - Rush Presbyterian - St. Luke's Medical Center, Chicago, Illinois
  - Children's Asthma Respiratory & Exercise Specialists, Glenview, Illinois
  - Cardinal Respiratory, PC, Springfield, Illinois
  - Clinical Research Center of Indiana, Indianapolis, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Consultants in Pulmonary Medicine, Olathe, Kansas
  - Heartland Research Associates, Wichita, Kansas
  - Northshore Medical Research, Covington, Louisiana
  - Institute for Asthma & Allergy, PC, Wheaton, Maryland
  - Center for Clinical Research, Taunton, Massachusetts
  - Henry Ford Hospital & Medical Centers, Detroit, Michigan
  - Hurley Child and Adolescent Asthma Center, Flint, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - Allergy, Asthma, Immunology Services, LLC, Jefferson City, Missouri
  - Midwest Chest Consultants, PC, Saint Charles, Missouri
  - Washington University School of Medicine, Division of Allergy & Immunology, St Louis, Missouri
  - Montana Medical Research, LLC, Missoula, Montana
  - Allergy, Asthma & Immunology Associates, PC, Lincoln, Nebraska
  - Heartland Clinical Research Inc., Omaha, Nebraska
  - Office of Meera Dewan, MD, Omaha, Nebraska
  - Delaware Valley Institute for Clinical Research, Cherry Hill, New Jersey
  - Clinical Research Center of Allergy & Asthma Consultants, Tinton Falls, New Jersey
  - Lovelace Scientific Resources, Albuquerque, New Mexico
  - Allergy & Asthma of Northern NM, Los Alamos, New Mexico
  - Pulmonary Medical Research of NY, Bay Shore, New York
  - Asthma & Allergy Associates, PC, Cortland, New York
  - Office of Michael Marcus, MD, Staten Island, New York
  - Office of Richard Castaldo, Tonawanda, New York
  - Regional Allergy & Asthma Consultants, Asheville, North Carolina
  - Charlotte Lung & Health Center, Charlotte, North Carolina
  - Neem Research Group, Inc., Charlotte, North Carolina
  - Cornerstone Research Care, High Point, North Carolina
  - Carolina MedTrials, LLC, Winston-Salem, North Carolina
  - Allergy & Asthma Care Center, Fargo, North Dakota
  - Sterling Research Group, Cincinnati, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Optimed Research LLC, Columbus, Ohio
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Allergy, Asthma and Dermatology Research Center, Lake Oswego, Oregon
  - Medford Medical Clinic, LLP, Medford, Oregon
  - Bellevue Pediatric Associates, Bellevue, Pennsylvania
  - Valley Clinical Research Center, Easton, Pennsylvania
  - Allergy & Asthma Research of NJ, Inc., Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Advanced Clinical Concepts, Shillington, Pennsylvania
  - Neem Research Group of Charleston, Charleston, South Carolina
  - Neem Research Group Inc., Columbia, South Carolina
  - Allergic Disease & Asthma Center, PA, Greenville, South Carolina
  - Asthma Institute, Chattanooga, Tennessee
  - The Allergy Associates, Knoxville, Tennessee
  - Office of Constantine Saadeh, Amarillo, Texas
  - Allergy & Asthma Clinical of Central Texas, Austin, Texas
  - UTX Medical, Galveston, Texas
  - Breco Research, Houston, Texas
  - Breath of Life Research Institute, Houston, Texas
  - Clinical Trials of North Houston, Houston, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Lung Diagnostics, San Antonio, Texas
  - Hampton Roads Center for Clinical Research, Norfolk, Virginia
  - Pulmonary Associates of Richmond Inc., Richmond, Virginia
  - Virginia Adult & Pediatric Allergy & Asthma PC, Richmond, Virginia
  - National Clinical Research, Richmond, Virginia
  - The Physician's Clinic of Spokane, Spokane, Washington
  - Allergy, Asthma, and Sinus Center F.C., Greenfield, Wisconsin
  - Milwaukee Medical Clinic, Milwaukee, Wisconsin
  - Allergic Diseases, S.C., West Allis, Wisconsin
- Canada (5):
  - Trial Management Group, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Clinical Research Group, Mississauga, Ontario
  - Niagara Clinical Research, Inc., Niagara Falls, Ontario
  - Primary Care Lung Clinic, Toronto, Ontario